CLINICAL TRIAL: NCT05913193
Title: High Calorie and High Protein Diabetes-specific Oral Nutritional Supplement in Type 2 Diabetes Subjects With or at Risk of Malnutrition in Real-life Setting: A Post-marketing Observational Study (PMO)
Brief Title: Oral Nutritional Supplement in Type 2 Diabetes Subjects With or at Risk of Malnutrition
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA31
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Malnutrition; Diabetes
MeSH Terms: conditions — Malnutrition; Diabetes Mellitus | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral Nutritional Supplement (ONS) Group: 2 servings per day as per standard of care during the study period
  Interventions: Other: Oral Nutritional Supplement (ONS)

INTERVENTIONS:
Other: Oral Nutritional Supplement (ONS) — Diabetes specific oral nutritional supplement

SUMMARY:
This multicenter, prospective study will evaluate the use of a nutritional support program including an oral diabetes-specific nutritional supplement consumed twice a day on the nutritional status of patients with T2D with or at risk of malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes on treatment with one or more oral antidiabetics/insulin and constant dose for at least 2 months
* Has HbA1c < 9.0% based on recent (30 days prior to Baseline visit) laboratory value or analysis of blood sample obtained at Baseline Visit
* Adult population with age ≥30 years
* Willing to follow the protocol as described
* Voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to any participation in the study to allow their data to be collected
* Subject is under the care of a health care professional for malnutrition, or is at risk for malnutrition (MUST≥1), and has recently (within the last 7 days prior to participating in this study) been prescribed study oral nutritional supplement (2 servings/day) by their health care professional

Exclusion Criteria:

* History of T2D longer than 30 years
* History of diabetic ketoacidosis and or hyperosmolar hyperglycemic state (HHS)
* If on thyroid medication or hormone replacement therapy, has not been on a constant dosage for at least 2 months prior to Baseline Visit
* History of metabolic/endocrine (other than diabetes), hepatic (AST/ALT 3 times the upper normal limit), or significant renal disease (GFR < 60 ml/min/1.73m2)
* History of heart failure (> class II)
* Follows a non-typical eating pattern, such as very low carbohydrate diet (e.g., Atkins diet, ketogenic diet, high protein diet), strict vegetarianism (e.g., no meat, dairy, eggs).
* Is pregnant as confirmed via urine pregnancy test, attempting to conceive or not willing and able to practice birth control during the study duration
* Has current infection (requiring medication or which might be expected to require hospitalization); has had inpatient surgery, or corticosteroid treatment (excluding topical creams) in the last 3 months or antibiotics in the last 3 weeks prior to Baseline Visit.
* Has an active malignancy
* Known to be allergic or intolerant to any ingredient found in the study products
* Taking any medications, herbals, or dietary supplements, other than allowed medications, during the past 4 weeks that could profoundly affect (in the opinion of the PI or study physician) blood glucose or appetite modifying medications (examples include orlistat, contrive, incretins, cannabis).
* Has known dementia, eating disorders, history of significant neurological or psychiatric disorder, or any other psychological condition that may interfere with study product consumption AND does not have a caregiver who can assist them with adherence to the study protocol
* Participant in a concomitant AN trial or trial of a nonregistered drug (or is within the 30 days follow-up period for such a trial) or that otherwise conflicts with this study unless otherwise approved by Abbott Nutrition.
* Patient is receiving any other oral supplement with HMB for nutritional management in the last 7 days

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with type 2 diabetes receiving an oral nutritional supplement as standard of care will be recruited from the investigator's community population.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Nutritional status risk by MUST | Baseline to Day 90
  Change in status as assessed by the Malnutrition Universal Screening Tool (MUST); Higher score indicates greater risk of malnutrition

SECONDARY OUTCOMES:
Blood Glycemic Measurement | Baseline to Day 90
  Change in glycemic control markers where lower levels are associated with improved control
Handgrip Strength | Baseline to Day 90
  Change in handgrip as measured in kg
Chair Stand Test | Baseline to Day 90
  Change in test score where higher number of times completed is more favorable
Body Composition | Baseline to Day 90
  Change in body composition where increased fat free mass is more favorable
EQ-5D Quality of Life | Baseline to Day 90
  Participant assessed 5 Domains; Each Domain scored from 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Diabetes Distress Scale | Baseline to Day 90
  Participant assessed 29 questions rated from 1 to 5 where higher number if less favorable
Subjective Global Assessment | Baseline to Day 90
  Healthcare Professional completed assessment of 4 components resulting in score where A = Well Nourished, B = Moderately Malnourished, and C = Severely Malnourished
Global Leadership Initiative on Malnutrition (GLIM) Diagnosis of Malnutrition | Baseline to Day 90
  Change in GLIM as calculated from MUST malnutrition risk and Phenotypic and Etiological Criteria

OTHER OUTCOMES:
Study Product Compliance | Baseline to Day 90
  Participant completed daily record of nutritional support program
Participant Satisfaction Survey | Day 90 or Early Exit
  Participant assessed 4 questions related to the nutritional support program scored from 1 to 10 where higher number is more favorable
Health Care Professional Satisfaction Survey | Day 90 or Early Exit
  Health Care Professional assessed 8 questions related to each Participant's study experience
Medication Usage | Baseline to Day 60 to Day 90
  Medications prescribed for glucose or appetite control
Body Mass Index | Baseline to Day 90
  As calculated from Height and Weight
Calf Circumference | Baseline to Day 90
  Measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: German Guzman, MD, Study Chair — Abbott
Locations (17):
- Spain (17):
  - Hospital Reina Sophia, Córdoba, Cordoba
  - Hospital Especialidades Virgen De La Victoria, Málaga, Malaga
  - Hospital Regional Malaga, Málaga, Malaga
  - Hospital Universitario Basurto, Bilbao
  - Hospital Uni. Puerta Del Mar, Cadiz
  - Hospital Virgen De Las Nieves, Granda
  - Hospital Juhn Romon Jimenez, Huelva
  - Hospital Universitario Jaen, Jaén
  - Complejo Hospitalario Universitario Insular-Materno infantil, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Virgen Del Rocio, Seville
  - Hospital Clinico Valencia, Valencia
  - Hospital La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No